CLINICAL TRIAL: NCT02776995
Title: Tumor Monitoring Using Thermography During Radiation Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Dr. Merav Ben-David, Medical and Radiation Oncologist, Head of Breast Radioation Unit, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1216-14-SMC
Record Dates: First submitted 2016-05-10; First posted 2016-05-19 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Malignancy
MeSH Terms: conditions — Neoplasms | interventions — Thermography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients undergoing radiation (Other): In this study, patients undergoing radiation treatment will undergo thermography imaging during radiation treatment course. Patients will be evaluated with thermography imaging every 5 fraction of radiation, starting prior to the first radiation treatment, periodically, until the end of radiation therapy (a period of several weeks).
  Interventions: Other: Thermography imaging

INTERVENTIONS:
Other: Thermography imaging — Thermography imaging of the treated - irradiated body area.

SUMMARY:
This research aims to investigate the correlation between tumor temperature difference and biological factors, such as size, metabolism, treatment response, and tumor aggressiveness.

In addition, normal tissue response to adjuvant radiation therapy in treated organs following surgery, will be evaluated.

DETAILED DESCRIPTION:
During radiation session, the investigators would evaluate the changes that will be detected by thermal imaging and correlate them with visible side effects as well as with known tumor biology factors and skin-tumor distance.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* will undergo radiation therapy for palliation or curative intent due to cancer, biopsy proven

Exclusion Criteria:

* not eligible to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-11; Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Measurement of IR : Infra-Red radiation emitted at wavelengths 0.8-1nm | Before the first fraction of radiation and every 5 fraction until the end of radiation therapy, approximately 4-5 weeks.
  Mathematical analysis of the thermic image

SECONDARY OUTCOMES:
Dermal side effects during radiation therapy using CTCAE v4.0 | Before the first fraction of radiation and every 5 fraction until the end of radiation therapy, approximately 4-5 weeks.
  Clinical assesment of the side effects by physician.
US/CT scans | The tumor size in cubic cm will be mesured prior to first fraction of radiation, and 2 weeks following the end of radiation session. Time for final evaluation: approximately 6-7 weeks.
  The tumor size will be measures to evaluate the efficacy of the radiation treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Merav Ben-David, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Merav Ben David, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No